CLINICAL TRIAL: NCT05853380
Title: A Multi-Center Prospective Open Label Study of a Web-based Application for Pulse Rate in Adult Patients
Status: Completed | Type: Observational
Sponsor: Mindset Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: IVC-400-006
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-06

CONDITIONS: Vital Sign Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Informed Vital Core App — All subjects assigned to a single arm, pulse rate measurement will be collected, calculated, and displayed on the web based application. A conventional ECG device will also be used to collect and display the heart rate at the same time. If additional consent is obtained subjects may provide blood pressure and SpO2 measurements for the web based application.

SUMMARY:
Evaluating the Accuracy of a Web-Based Application - Vital Sign Measurement Platform Description This single-arm cohort, open-label, and multi-center study is designed to evaluate the accuracy of a web-based application designed for measurements of vital signs including pulse rate (PR). It is hypothesized that the accuracy of the App is non-inferior to the accuracy of an FDA-cleared/approved vital sign monitoring device (reference device).

ELIGIBILITY:
Inclusion Criteria:

* Subjects 22 -85 years of age
* Subjects willing to sign the Informed Consent Form and comply with the protocol

Exclusion Criteria

* Subjects required to wear mask or bandage that obstructs forehead, cheeks, or chin
* Refusal to remove makeup , sunscreen, lotion, clothing, or items obstructing the face for the duration of measurement
* Presence of facial tattoos, large birthmarks, or other skin alterations (scars, hemangiomas, vitiligo) on upper cheeks (cheekbone) or forehead of the subject
* Condition that does not allow the subject to remain still for 60 seconds at a time
* Subjects with cardiac arrhythmia
* Any known medical condition which may result in an inaccurate measurement using the reference device
* Subjects with the inability to complete an ECG.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit subjects from clinics and hospitals and the general public. Enrollment of 85 subjects with an age range of 22-85 years of age with a wide range of skin tone categorization per the Fitzpatrick Scale ranging from 1-6.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Lubelski, MD, Principal Investigator — Mindset Medical
Locations (6):
- United States (6):
  - Velocity Clinical Research, Mobile, Alabama
  - Velocity Clinical Research, La Mesa, California
  - Velocity Clinical Research, Meridian, Idaho
  - Velocity Clinical Research, Cleveland, Ohio
  - Velocity Clinical Research, Columbia, South Carolina
  - Velocity Clinical Research, Cedar Park, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited subjects from clinics, hospitals, and the general public. The study was conducted in the United States.
Groups:
- Single Arm: Open Label, Single Group Assignment
Period: Overall Study
Arm/Group | Single Arm
Started | 86
Completed | 82
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Intent to Measure
Arm/Group | Single Arm
Number analyzed (Participants) | 82
Age, Continuous [Mean (Full Range); unit: Years] | 48.7 [22 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 32
  White | 41
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 82
IVC App Pulse Rate [Median (Inter-Quartile Range); unit: Beats per Minute] — ECG Heart Rate (beats per minute) Population: ECG HR is reported for the 69 subjects with comparator data.
  Beats per Minute
    number analyzed (Participants) | 69
    (all) | 69.0 [63 to 77]
IVC App Report Rate [Count of Participants; unit: Participants] — Population: IVC App successfully reported the Pulse Rate for 69 of 82 subjects
  Participants | 69

OUTCOME MEASURES:

1. Primary Outcome: Pulse Rate Accuracy
Description: The primary endpoint is a comparison to an FDA-cleared reference device to establish that PR measured with the IVC App is accurate.
Time Frame: 120 seconds
Population: Intent to Capture
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 82
Participants | 67
Statistical Analysis 1: Comparison: Single Arm; Subjects with simultaneously collected HR and PR comparator data were assigned to the comparison group; Test type: Other — The primary outcome was considered successful if the bootstrapped upper 95% confidence interval on the RMSD was < 3.0. Power was assessed by bootstrapping 95% confidence intervals at different n sizes on a product development population; RMSD = 0.77, 95% CI 2-sided [0.67 to 0.87]; The upper 95% confidence interval on the RMSD was 0.87, meeting the significance threshold of < 3.0. The study tested hypothesis of accuracy < 3.0 RMSD by showing the upper 95% confidence interval on the RMSD was < 3.0. The upper 95% confidence interval on the RMSD was 0.87, meeting the target threshold of < 3.0

ADVERSE EVENTS:
Time Frame: 120 seconds
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT05853380/Prot_SAP_000.pdf